CLINICAL TRIAL: NCT00142480
Title: Phase II Study of Capecitabine, Oxaliplatin, Bevacizumab and Radiation Therapy in Biliary Tract and Gallbladder Cancer
Brief Title: Capecitabine, Oxaliplatin, Bevacizumab and Radiation Therapy in Patients With Biliary Tract and Gallbladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Genentech, Inc. (Industry); Sanofi-Synthelabo (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Andrew X. Zhu, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-144
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Biliary Tract Cancer; Gallbladder Adenocarcinoma
Keywords: locally advanced biliary adenocarcinoma; unresectable biliary adenocarcinoma; gallbladder adenocarcinoma; capecitabine; oxaliplatin; bevacizumab; Biliary tract adenocarcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Capecitabine; Oxaliplatin; Bevacizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine, Oxaliplatin, Bevacizumab (Experimental): There are two phases of study treatment. Phase I includes all patients and will last 6 weeks. During this phase, oxaliplatin will be given intravenously (IV) on days 1, 8, 22, and 29; bevacizumab will be given IV on days 1, 15, and 29; capecitabine will be administered orally on days 1-14 and 22-35. Radiation therapy will be given once daily for 5 days (Monday-Friday) per week for a total of 28 treatments. Phase II has two groups: 1) patients who had tumors removed prior to entering study and 2) patients who entered the study with advanced disease. Patients who had their tumors removed prior to entering the study will be treated with the above 6-week regimen twice for a total of 12 weeks of treatment. Patients who were unresectable prior to entering the study but then were deemed resectable after treatment on trial will undergo resection. Following surgical recovery (8-10 weeks) they will be treated again with the above 6-week regimen twice for a total of 12 weeks of treatment.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Bevacizumab; Procedure: Radiation therapy

INTERVENTIONS:
Drug: Capecitabine — Given orally for 14 consecutive days (days 1-14) followed by a week of no capecitabine then another week of 14 consecutive days (days 21-28).
Drug: Oxaliplatin — Given intravenously once weekly during weeks 1, 2, 4 and 5 on days 1, 8, 22 and 29
Drug: Bevacizumab — Given intravenously every two weeks during weeks 1, 3 and 5 on days 1, 15 and 29.
Procedure: Radiation therapy — Once daily for 5 days (Monday through Friday) for a total of 28 treatments.

SUMMARY:
The main purpose of this study is to test the safety and effectiveness of oxaliplatin, bevacizumab, and capecitabine given in combination with radiation therapy to see what effects (good or bad) they have on patients with biliary tract and gallbladder cancer.

DETAILED DESCRIPTION:
There are two phases of study treatment. The first phase is for all patients and will last about 6 weeks. During this phase, oxaliplatin will be given intravenously once a week during weeks 1, 2, 4, and 5 on days 1, 8, 22, and 29; bevacizumab will be given intravenously once every 2 weeks during weeks 1, 3, and 5 on days 1, 15, and 29; capecitabine will be administered orally for 14 consecutive days (days 1-14), then a week of no capecitabine, followed by another 14 days of capecitabine (days 22-35).

Radiation therapy will be given once daily for 5 days (Monday-Friday) per week for a total of 28 treatments.

During this first phase of the study the following tests will be performed weekly: physical exam, vital signs, medical history, blood tests and urine tests.

After the first phase is finished patients will wait 4 weeks then have a CT scan, MRCP, blood tests and a physical exam to evaluate the status of the disease.

Phase two of the study is broken up into two groups: 1) patients who had tumors removed prior to entering study and 2) patients who entered the study with advanced disease.

If the patients had tumors removed prior to entering the study, they will be treated again with all 3 study drugs but no radiation over a 6-week period as they did earlier in the study. This 6-week regimen will be repeated twice for a total of 12 weeks of treatment.

Patients with advanced disease that could not be removed by surgery when they first entered the study but the evaluation tests after the first phase show the tumor has responded (reduced in size) and can now be resected, will have surgery to remove the tumors.

Following surgical recovery (8-10 weeks) they will be treated again with all 3 of the study drugs but no radiation over a 6-week period as they did earlier in the study. This 6-week regimen will be repeated twice for a total of 12 weeks of study treatment.

If the evaluation tests show that the patients' cancer has remained stable (not gotten worse or better) they will be treated again with all three study drugs but no radiation over a 6-week period as they did earlier in the study. This 6-week regimen will be repeated twice for a total of 12 weeks of study treatment.

During the additional 12 weeks of study treatment a physical exam, vital signs, medical history, blood testing and urine testing will be performed once every 3 weeks.

At the end of study treatment the following evaluations will be performed: physical exam, vital signs, blood work, CT scan of the chest and abdomen, MRCP, and tumor measurements by CT scans. These evaluations will be repeated every 3 months thereafter.

Patients will be removed from the study if their disease worsens or there are unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced unresectable biliary tract or gallbladder adenocarcinoma
* Patients with resected biliary tract or gallbladder adenocarcinoma who have residual tumor left will also be eligible.
* > 4 weeks since time of major surgery
* > 2 weeks since time of minor surgery
* > 4 weeks since time of major radiotherapy for other malignancy
* > 4 weeks since participation in any investigational drug study
* > 1 year since treatment for other carcinomas, except cured non-melanoma skin and treated in-situ cervical cancer
* 18 years of age or older
* ECOG performance status of 0-2
* Life expectancy > 12 weeks
* Absolute neutrophil count (ANC) > 1,500/mm3
* Hemoglobin > 9.0 gm/dl
* Platelets > 100,000/mm3
* SGOT < 5 x upper limits of normal (ULN)
* Total bilirubin < 2.5 mg/dl
* Creatinine clearance > 50 ml/min

Exclusion Criteria:

* Prior chemotherapy or radiation therapy for biliary tract or gallbladder cancer
* Peripheral neuropathy of grade 2 or greater
* Unstable angina
* Symptomatic congestive heart failure
* Myocardial infarction < 12 months prior to registration
* New York Heart Association classification III or IV
* Active or uncontrolled infection
* Known existing uncontrolled coagulopathy
* Malabsorption syndrome or lack of integrity of the upper gastrointestinal (GI) tract
* Prior unanticipated severe reaction to fluoropyrimidine therapy or known sensitivity to 5-fluorouracil, or known dihydropyrimidine dehydrogenase (DPD) deficiency
* Known brain metastases or carcinomatous meningitis
* Pregnant or lactating women
* Serious, non-healing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-12; Primary Completion 2007-07 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To determine the progression free survival rate at one year for locally advanced, or resected with positive margins, biliary tract and gallbladder cancer patients | 3 years

SECONDARY OUTCOMES:
To evaluate the safety of the combination capecitabine, oxaliplatin, bevacizumab in patients with biliary tract and gallbladder cancer | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zhu, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts